CLINICAL TRIAL: NCT02481596
Title: Family-Focused Mobile Health Intervention: Targeting Family Behaviors to Improve Type 2 Diabetes Management Among Adults
Brief Title: FAMS Mobile Health Intervention for Diabetes Self-care Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Lindsay Mayberry, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 140562_A
Record Dates: First submitted 2015-06-23; First posted 2015-06-25 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: family; support; diet; exercise; social
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Masking Description: The outcomes assessor for the primary outcome for the larger trial (NCT02409329) was blinded, but outcomes assessors for these outcomes were not.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- REACH + FAMS (Experimental): Participants will receive FAMS components (monthly phone coaching and text messages supporting a goal set in coaching, plus the option to invite a family member/support person to receive text messages) for six months.
  All participants will receive text messages advising how to access their study A1c test results, quarterly newsletters on healthy living with diabetes, and have access to a Helpline for study- and diabetes medication-related questions.
  Interventions: Behavioral: REACH + FAMS; Behavioral: REACH; Behavioral: Helpline & A1c results
- REACH (Experimental): Participants will receive REACH text messages (individual-focused text messaging tailored to user's individual barriers to adherence, messages assessing medication adherence with feedback, and targeted to address other self-care behaviors).
  All participants will receive text messages advising how to access their study A1c test results, quarterly newsletters on healthy living with diabetes, and have access to a Helpline for study- and diabetes medication-related questions.
  Interventions: Behavioral: REACH; Behavioral: Helpline & A1c results
- Helpline & A1c results (Active Comparator): Participants assigned to the control group will complete measures at each time point and maintain care as usual (i.e., medical treatment and physician monitoring).
  All participants will receive text messages advising how to access their study A1c test results, quarterly newsletters on healthy living with diabetes, and have access to a Helpline for study- and diabetes medication-related questions.
  Interventions: Behavioral: Helpline & A1c results

INTERVENTIONS:
Behavioral: REACH + FAMS — The intervention consists of REACH individual-focused text messaging, plus family-focused phone coaching sessions, goal-focused text messaging, and the option to invite a family member/support person to receive text messages.
  Other Names: Family-focused intervention
  Arms: REACH + FAMS
Behavioral: REACH — The intervention consists of daily text messaging tailored to user's individual barriers to medication adherence, plus text messaging targeting other self-care behaviors (see NCT02409329).
  Other Names: NCT02409329
  Arms: REACH; REACH + FAMS
Behavioral: Helpline & A1c results — Participants complete all study assessments, receive text messages advising how to access study A1c results, and have access to a helpline for study- or diabetes medication-related questions.

SUMMARY:
This study evaluates a family-focused mobile phone-delivered intervention, called FAMS (Family-focused Add-on for Motivating Self-care), in supporting adults with type 2 diabetes in their self-management relative to a control group. The goal of this study is to ascertain if family-focused content delivered to the patient can improve the patients' family support for diabetes self-care, self-efficacy, and adherence to diet and exercise recommendations.

DETAILED DESCRIPTION:
Family members perform diabetes-specific behaviors that are helpful and/or harmful to the adult managing type 2 diabetes. Family behaviors are strongly associated with patients' adherence to diet and exercise: supportive family behaviors with more adherence and harmful family behaviors with less adherence. This six-month intervention seeks to increase supportive and reduce harmful family behaviors, and to improve diabetes-related self-efficacy and adherence to diet and exercise recommendations among adult patients with content that can be delivered via basic mobile phones (i.e., phone calls and text messages).

FAMS components include:

* Six 20-30 minute coaching sessions with patient participants by phone focusing on helpful/unhelpful/desired family behaviors relevant to the patients' self-identified daily diet or exercise goal (occurs after enrollment and monthly for six months)
* Text messages to the patient to support him/her in meeting the identified daily goal (4 per week)
* The option to invite an adult support person to receive text messages (3 per week) encouraging the support person to discuss the patient's self-care goal to provide opportunities for the patient to practice skills discussed during phone coaching

This intervention evaluation is nested within a larger randomized controlled trial (RCT; see NCT02409329) which evaluates REACH, a text messaging intervention to improve participants' adherence to self-care and glycemic control. We will evaluate these interventions with a three arm trial. Participants will be randomized to receive REACH only, REACH+FAMS, or an active control. Participants assigned to REACH+FAMS will receive the above described components for the first six months of the trial, and then REACH only until the end of the trial. Analyses will examine outcomes of FAMS at 3 and 6 months.

ELIGIBILITY:
*Note: Criteria for patient participants is consistent with larger study (NCT02409329).

Inclusion Criteria:

* Adults aged 18 years and older
* Individuals who have received a diagnosis for type 2 diabetes mellitus
* Enrolled as a patient at a participating community health center
* Individuals currently being treated with oral and/or injectable diabetes medications

Exclusion Criteria:

* Non-English speakers
* Individuals who report they do not have a cell phone
* Individuals unwilling and/or not able to provide written informed consent
* Individuals with unintelligible speech (e.g., dysarthria)
* Individuals with a severe hearing or visual impairment
* Individuals who report a caregiver administers their diabetes medications
* Individuals who fail the cognitive screener administered during the baseline survey
* Individuals who cannot receive, read, and respond to a text after instruction from a trained research assistant

Support persons invited to receive text messages must meet following criteria:

Support Person Inclusion Criteria:

* Adults aged 18 years and older
* Identified by the patient as a part of their family (can be related biologically or legally, or be a close friend/roommate who participates in the patients' daily routine)

Support Person Exclusion Criteria:

* Non-English speakers (determined subjectively by a trained research assistant)
* Individuals who report they do not have a cell phone
* Individuals unwilling and/or not able to provide written informed consent
* Individuals with unintelligible speech (e.g., dysarthria) (determined subjectively by a trained research assistant)
* Individuals with a severe hearing or visual impairment (determined subjectively by a trained research assistant)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2016-05-23 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay S Mayberry, MS, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Federally Qualified Health Centers & Vanderbilt Primary Care Clinics, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data collected during the trial will be de-identified and made available following publication of the 15-month trial results (see NCT02409329) to researchers who provide a methodologically sound proposal.
Supporting Information: Study Protocol
Time Frame: Beginning 6 months after final trial results publication. No end date.
Access Criteria: Approval of a proposal by the study PI.

REFERENCES:
- [Background] Mayberry LS, Berg CA, Harper KJ, Osborn CY. The Design, Usability, and Feasibility of a Family-Focused Diabetes Self-Care Support mHealth Intervention for Diverse, Low-Income Adults with Type 2 Diabetes. J Diabetes Res. 2016;2016:7586385. doi: 10.1155/2016/7586385. Epub 2016 Nov 7. PMID 27891524
- [Background] Nelson LA, Wallston KA, Kripalani S, Greevy RA Jr, Elasy TA, Bergner EM, Gentry CK, Mayberry LS. Mobile Phone Support for Diabetes Self-Care Among Diverse Adults: Protocol for a Three-Arm Randomized Controlled Trial. JMIR Res Protoc. 2018 Apr 10;7(4):e92. doi: 10.2196/resprot.9443. PMID 29636319
- [Derived] Mayberry LS, Berg CA, Greevy RA, Nelson LA, Bergner EM, Wallston KA, Harper KJ, Elasy TA. Mixed-Methods Randomized Evaluation of FAMS: A Mobile Phone-Delivered Intervention to Improve Family/Friend Involvement in Adults' Type 2 Diabetes Self-Care. Ann Behav Med. 2021 Mar 16;55(2):165-178. doi: 10.1093/abm/kaaa041. PMID 32706852

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 subjects were never reached for a required conversation prior to starting the text messaging program--they were withdrawn by the PI. 1 subject was withdrawn by the PI due to problematic behavior during enrollment.
Groups:
- REACH + FAMS: Participants will receive FAMS components (monthly phone coaching and text messages supporting a goal set in coaching, plus the option to invite a family member/support person to receive text messages) for six months.
  All participants will receive text messages advising how to access their study A1c test results, quarterly newsletters on healthy living with diabetes, and have access to a Helpline for study- and diabetes medication-related questions.
  REACH + FAMS: The intervention consists of REACH individual-focused text messaging, plus family-focused phone coaching sessions, goal-focused text messaging, and the option to invite a family member/support person to receive text messages.
- REACH: Participants will receive REACH text messages (individual-focused text messaging tailored to user's individual barriers to adherence, messages assessing medication adherence with feedback, and targeted to address other self-care behaviors).
  All participants will receive text messages advising how to access their study A1c test results, quarterly newsletters on healthy living with diabetes, and have access to a Helpline for study- and diabetes medication-related questions.
  REACH: The intervention consists of daily text messaging tailored to user's individual barriers to medication adherence, plus text messaging targeting other self-care behaviors (see NCT02409329).
  Helpline & A1c results: Participants complete all study assessments, receive text messages advising how to access study A1c results, and have access to a helpline for study- or diabetes medication-related questions.
- Helpline & A1c Results: Participants assigned to the control group will complete measures at each time point and maintain care as usual (i.e., medical treatment and physician monitoring).
  All participants will receive text messages advising how to access their study A1c test results, quarterly newsletters on healthy living with diabetes, and have access to a Helpline for study- and diabetes medication-related questions.
  Helpline & A1c results: Participants complete all study assessments, receive text messages advising how to access study A1c results, and have access to a helpline for study- or diabetes medication-related questions.
Period: Overall Study
Arm/Group | REACH + FAMS | REACH | Helpline & A1c Results
Started | 126 | 127 | 253
Completed | 123 | 126 | 245
Not Completed | 3 | 1 | 8

BASELINE CHARACTERISTICS:
Groups:
- REACH + FAMS: Participants will receive FAMS components (monthly phone coaching and text messages supporting goal set in coaching, plus the option to invite a support person to receive text messages) for six months.
  All participants will receive text messages advising how to access their study A1c test results, quarterly newsletters on healthy living with diabetes, and have access to a Helpline for study- and diabetes medication-related questions.
- Total: Total of all reporting groups
Arm/Group | REACH + FAMS | REACH | Helpline & A1c Results | Total
Number analyzed (Participants) | 126 | 127 | 253 | 506
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 97 | 109 | 206 | 412
  >=65 years | 29 | 18 | 47 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (10.2) | 55.8 (9.4) | 56.1 (9.4) | 55.9 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 70 | 135 | 274
  Male | 57 | 57 | 118 | 232
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 15 | 31
  Not Hispanic or Latino | 111 | 116 | 224 | 451
  Unknown or Not Reported | 7 | 3 | 14 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 3 | 4
  Asian | 2 | 3 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 49 | 51 | 98 | 198
  White | 63 | 64 | 128 | 255
  More than one race | 5 | 2 | 6 | 13
  Unknown or Not Reported | 6 | 6 | 15 | 27
Region of Enrollment [Number; unit: participants]
  United States | 126 | 127 | 253 | 506
Problem eating behaviors - Personal Diabetes Questionnaire [Median (Inter-Quartile Range); unit: units on a scale] — as measured by Personal Diabetes Questionnaire diet subscale Problem Eating Behavior (1=less problem eating behavior - better to 6=more problem eating behavior - worse)
  units on a scale | 3.3 [2.7 to 4.0] | 3.3 [2.3 to 4.0] | 3.3 [2.7 to 4.0] | 3.3 [2.7 to 4.0]
Use of dietary information - Personal Diabetes Questionnaire [Median (Inter-Quartile Range); unit: units on a scale] — as measured by Personal Diabetes Questionnaire diet subscale Use of Dietary Information for Decision Making (1=less use of information - worse to 6=more use of information - better)
  units on a scale | 2.7 [1.3 to 4.0] | 3.0 [1.0 to 4.7] | 2.7 [1.0 to 4.3] | 3.0 [1.0 to 4.3]
MET-minutes per week - International Physical Activity Questionnaire-short form [Median (Inter-Quartile Range); unit: MET-minutes per week] — metabolic equivalent minutes (MET-minutes) per week where more MET-minutes per week indicates more physical activity
  MET-minutes per week | 1158 [339 to 2655] | 1448 [520 to 3560] | 1299 [236 to 3492] | 1352 [386 to 3348]
Helpful involvement - Family and Friend Involvement in Adults' Diabetes [Median (Inter-Quartile Range); unit: units on a scale] — as measured by Family and Friend Involvement in Adults' Diabetes (FIAD) helpful involvement subscale ranging from 1= less frequent helpful involvement (worse) to 5=more frequent helpful involvement (better)
  units on a scale | 1.8 [1.2 to 2.3] | 1.6 [1.1 to 2.4] | 1.9 [1.2 to 2.6] | 1.8 [1.2 to 2.4]
Harmful involvement - Family and Friend Involvement in Adults' Diabetes [Median (Inter-Quartile Range); unit: units on a scale] — as measured by Family and Friend Involvement in Adults' Diabetes (FIAD) harmful involvement subscale ranging from 1= less frequent harmful involvement (better) to 5=more frequent harmful involvement (worse)
  units on a scale | 1.6 [1.3 to 2.1] | 1.6 [1.1 to 2.0] | 1.6 [1.4 to 2.0] | 1.6 [1.3 to 2.0]
Diabetes self-efficacy - Perceived Diabetes Self-Management Scale [Median (Inter-Quartile Range); unit: units on a scale] — as measured by scores on the Perceived Diabetes Self-Management Scale (4-item version) ranging from 4 = low self-efficacy (worse) to 20 = high self-efficacy (better)
  units on a scale | 14 [12 to 16] | 14 [12 to 17] | 14 [11 to 17] | 14 [11 to 16]

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Diet - Use of Dietary Information
Description: as measured by Personal Diabetes Questionnaire Use of Dietary Information for Decision Making (1=less use of information - worse to 6=more use of information - better)
Time Frame: 3 months, 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | REACH + FAMS | REACH | Helpline & A1c Results
Number analyzed (Participants) | 126 | 127 | 253
score on a scale
  3 months | 3.0 [1.7 to 4.3] | 3.3 [1.7 to 4.3] | 2.7 [1.0 to 4.0]
  6 months | 3.3 [2.0 to 4.3] | 3.3 [2.0 to 4.7] | 2.7 [1.3 to 4.3]
Statistical Analysis 1: Comparison: REACH + FAMS vs Helpline & A1c Results; 3 months. Multiply imputed data (m=20) using chained equations; Test type: Superiority; p = .045, Regression, Linear — Beta=.083. Threshold p<.05; Adjusted for baseline values with cubic splines (3 knots)
Statistical Analysis 2: Comparison: REACH + FAMS vs Helpline & A1c Results; 6 months. Multiply imputed data (m=20) using chained equations; Test type: Superiority; p = .006, Regression, Linear — Beta=.126. Threshold p<.05; Adjusted for baseline values with cubic splines (3 knots)

2. Primary Outcome: Adherence to Exercise
Description: as measured by International Physical Activity Questionnaire-Short form [metabolic equivalent minutes (MET-minutes) per week] where more MET-minutes per week indicates more physical activity
Time Frame: 3 months, 6 months
Measure: Median (Inter-Quartile Range); unit: MET-minutes per week
Arm/Group | REACH + FAMS | REACH | Helpline & A1c Results
Number analyzed (Participants) | 126 | 127 | 253
MET-minutes per week
  6 months | 1293 [558 to 3120] | 1000 [273 to 2240] | 1295 [438 to 2549]
  3 months | 1251 [510 to 2691] | 977 [248 to 2799] | 1187 [438 to 3210]
Statistical Analysis 1: Comparison: REACH + FAMS vs Helpline & A1c Results; 3 months. Multiply imputed data (m=20) using chained equations; Test type: Superiority; p = .518, Regression, Linear — Beta=.031. Threshold p<.05; Adjusted for baseline values with cubic splines (3 knots)
Statistical Analysis 2: Comparison: REACH + FAMS vs Helpline & A1c Results; 6 months. Multiply imputed data (m=20) using chained equations; Test type: Superiority; p = .092, Regression, Linear — Beta=.092. Threshold p<.05; Adjusted for baseline values with cubic splines (3 knots)

3. Primary Outcome: Adherence to Diet - Problem Eating Behavior
Description: as measured by Personal Diabetes Questionnaire diet subscale Problem Eating Behavior (1=less problem eating behavior - better to 6=more problem eating behavior - worse)
Time Frame: 3 months, 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | REACH + FAMS | REACH | Helpline & A1c Results
Number analyzed (Participants) | 126 | 127 | 253
score on a scale
  3 months | 3.3 [2.7 to 3.7] | 3.0 [2.3 to 3.7] | 3.0 [2.7 to 4.0]
  6 months | 3.3 [2.7 to 3.7] | 3.0 [2.3 to 3.7] | 3.0 [2.7 to 4.0]
Statistical Analysis 1: Comparison: REACH + FAMS vs Helpline & A1c Results; 3 months. Multiply imputed data (m=20) using chained equations; Test type: Superiority; p = .53, Regression, Linear — Beta=-.027. Threshold p<.05; Adjusted for baseline values with cubic splines (3 knots)
Statistical Analysis 2: Comparison: REACH + FAMS vs Helpline & A1c Results; 6 months. Multiply imputed data (m=20) using chained equations; Test type: Superiority; p = .41, Regression, Linear — Beta=-.037. Threshold p<.05; Adjusted for baseline values with cubic splines (3 knots)

4. Secondary Outcome: Supportive Family Behaviors
Description: as measured by Family and Friend Involvement in Adults' Diabetes (FIAD) helpful involvement subscale ranging from 1= less frequent helpful involvement (worse) to 5=more frequent helpful involvement (better)
Time Frame: 3 months, 6 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | REACH + FAMS | REACH | Helpline & A1c Results
Number analyzed (Participants) | 126 | 127 | 253
units on a scale
  3 months | 1.8 [1.4 to 2.7] | 1.6 [1.1 to 2.3] | 1.8 [1.2 to 2.6]
  6 months | 1.8 [1.3 to 2.7] | 1.6 [1.0 to 2.4] | 1.7 [1.2 to 2.4]
Statistical Analysis 1: Comparison: REACH + FAMS vs Helpline & A1c Results; 3 months. Multiply imputed data (m=20) using chained equations; Test type: Superiority; p = .024, Regression, Linear — Beta=.088. Threshold p<.05; Adjusted for baseline values with cubic splines (3 knots); also adjusted for harmful involvement subscale of FIAD due to suppression effect
Statistical Analysis 2: Comparison: REACH + FAMS vs Helpline & A1c Results; 6 months. Multiply imputed data (m=20) using chained equations; Test type: Superiority; p = .003, Regression, Linear — Beta=.128. Threshold p<.05; [statistical method as in outcome 4, analysis 1]

5. Secondary Outcome: Obstructive Family Behaviors
Description: as measured by Family and Friend Involvement in Adults' Diabetes (FIAD) harmful involvement subscale ranging from 1= less frequent harmful involvement (better) to 5=more frequent harmful involvement (worse)
Time Frame: 3 months, 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | REACH + FAMS | REACH | Helpline & A1c Results
Number analyzed (Participants) | 126 | 127 | 253
score on a scale
  3 months | 1.4 [1.1 to 1.9] | 1.4 [1.1 to 1.9] | 1.6 [1.1 to 2.0]
  6 months | 1.3 [1.0 to 1.9] | 1.4 [1.1 to 1.7] | 1.4 [1.1 to 1.9]
Statistical Analysis 1: Comparison: REACH + FAMS vs Helpline & A1c Results; 3 months. Multiply imputed data (m=20) using chained equations; Test type: Superiority; p = .001, Regression, Linear — Beta=-.133. Threshold p<.05; Adjusted for baseline values with cubic splines (3 knots); also adjusted for helpful involvement subscale of FIAD due to suppression effect
Statistical Analysis 2: Comparison: REACH + FAMS vs Helpline & A1c Results; 6 months. Multiply imputed data (m=20) using chained equations; Test type: Superiority; p = .012, Regression, Linear — Beta=-.115. Threshold p<.05; [statistical method as in outcome 5, analysis 1]

6. Secondary Outcome: Diabetes Self-efficacy
Description: as measured by scores on the Perceived Diabetes Self-Management Scale (4-item version) ranging from 4 = low self-efficacy (worse) to 20 = high self-efficacy (better)
Time Frame: 3 months, 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | REACH + FAMS | REACH | Helpline & A1c Results
Number analyzed (Participants) | 126 | 127 | 253
score on a scale
  3 months | 14 [12 to 17] | 15 [13 to 18] | 14 [11 to 16]
  6 months | 15 [12 to 17.5] | 15 [12 to 18] | 14 [12 to 16]
Statistical Analysis 1: Comparison: REACH + FAMS vs Helpline & A1c Results; 3 months. Multiply imputed data (m=20) using chained equations; Test type: Superiority; p = .015, Regression, Linear — Beta=.114. Threshold p<.05; Adjusted for baseline values with cubic splines (3 knots)
Statistical Analysis 2: Comparison: REACH + FAMS vs Helpline & A1c Results; 6 months. Multiply imputed data (m=20) using chained equations; Test type: Superiority; p = .034, Regression, Linear — Beta=.101. Threshold p<.05; Adjusted for baseline values with cubic splines (3 knots)

ADVERSE EVENTS:
Time Frame: We followed participants for 6 months of study participation, lasting from recruitment start May 2016 until the last participant completed 6-month follow-up in July 2018.
Arm/Group | REACH + FAMS | REACH | Helpline & A1c Results
All-Cause Mortality (participants affected / at risk) | 0/126 | 1/127 | 2/253
Serious Adverse Events (participants affected / at risk) | 0/126 | 0/127 | 0/253
Other Adverse Events (participants affected / at risk) | 0/126 | 0/127 | 0/253

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/96/NCT02481596/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/96/NCT02481596/SAP_001.pdf